CLINICAL TRIAL: NCT04403646
Title: Efficacy of Tannin Specific Natural Extract for Coronavirus Disease (COVID-19): Randomized Controlled Trial
Brief Title: Tannin Specific Natural Extract for COVID-19 Infection
Acronym: TanCOVID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low rate of covid patients
Sponsor: Hospital de Clinicas José de San Martín (Other)
Collaborators: SILVATEAM (Unknown)
Responsible Party: Principal Investigator, Maria Marta Piskorz, Neurogastroenterologist at Hospital de Clinicas, Principal Investigator, Hospital de Clinicas José de San Martín
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HCJSM-20-005
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: COVID-19; SARS-CoV 2; Coronavirus Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TREATED (Experimental): Participants will receive a supply of 28 -- 390 mg ARBOX capsules for 14 days. Patients will be supplemented with 2 capsules of ARBOX per day and standard therapy.
  Standard treatment includes: Antipyretics or Lopinavir / Ritonavir, Azithromycin and Hydroxychloroquine, as appropriate (treatment currently recommended by the department of Infectious Diseases of the Hospital de Clínicas that could undergo to modifications). In addition, if necessary: supplemental O2, non-invasive ventilation, antibiotic therapy.
  Interventions: Dietary Supplement: ARBOX
- CONTROL (Placebo Comparator): Participants will receive placebo supply for 14 days. The placebo will be administrated with the identical dose as described for the test product.
  Beside patients will receive the standard theraphy, which includes Antipyretics or Lopinavir / Ritonavir, Azithromycin and Hydroxychloroquine, as appropriate (treatment currently recommended by the department of Infectious Diseases of the Hospital de Clínicas that could undergo to modifications). In addition, if necessary: supplemental O2, non-invasive ventilation, antibiotic therapy.
  Interventions: Other: PLACEBO

INTERVENTIONS:
Dietary Supplement: ARBOX — dry extract of polyphenols (tannins) form quebracho and chestnut 240 mg, B12 vitamin 0.72 µg
  Arms: TREATED
Other: PLACEBO — Matching placebo, twice-daily administration BID as described for the test product, identical number of tablets as given for ARBOX
  Arms: CONTROL

SUMMARY:
There is an urgent need to evaluate interventions that could be effective against the infection with SARS-CoV 2. Tannins based wood extracts are an inexpensive and safe product with protective effect in both bacterial and viral infections likely due to its anti- inflammatory, anti-oxidative effects and their modulation of the intestinal microbiota. This randomized controlled trial seeks to evaluate the efficacy of the tannins based dietary supplement ARBOX in positive COVID-19 patients.

DETAILED DESCRIPTION:
The epidemic of 2019 novel coronavirus (causing the disease Covid-19) has expanded from Wuhan throughout China and is being exported to a growing number of countries, some of which have seen onward transmission. COVID-19 caused clusters of severe respiratory illness and was associated with 2% mortality. There is currently no vaccine and no specific antiviral treatment recommended for COVID-19. About 20% of the patients were severe and the mainstay of clinical management is largely symptomatic treatment, with organ support in intensive care for seriously ill patients. Therefore, it is urgent to find a safe and effective therapeutic approach to COVID-19.

Tannins have been shown to have antioxidant, anti-inflammatory, antimicrobial properties and a regulatory effect on the gastrointestinal metabolism.

The investigators will realize a prospective, double-blind, randomized trial to assess the effect of treatment with a dietary supplement (ARBOX), a molecular complex of quebracho and chestnut tannins extract and Vit B12, compared with placebo. 140 COVID-19 patients will be recruited in a single center in Buenos Aires Argentina. 70 patients will receive conventional treatment plus ARBOX (treated group) and 70 patients will receive conventional treatment plus placebo (control group). The effects will be evaluated during the 28 days follow up. The primary end point will be the time of discharge from the hospital. A panel of 27 cytokines level, intestinal microbiota composition and its metabolites will be assessed at day 1 and 14.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age hospitalized in the general hospitalization room, who meet the definition of "Confirmed case COVID-19" (https://www.argentina.gob.ar/salud/coronavirus-COVID-19/definicion -of-case)

Exclusion Criteria:

* Pregnancy
* Lactancy
* Hypersensitivity to polyphenols
* Patients unable to receive oral medication (severe cognitive impairment, assisted ventilation, impaired state of consciousness)
* Lack of consent
* Participation in any other interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Time to hospital discharge | Throughout the Study (Day 0 to Day 28)
  defined as the time from first dose of polyphenol extract to hospital discharge

SECONDARY OUTCOMES:
28-day all-cause mortality | Throughout the Study (Day 0 to Day 28)
  proportion
invasive ventilation on day 28 | Throughout the Study (Day 0 to Day 28)
  proportion
Difference in Pro and antiinflammatory citoquine levels | day 1-14
  mean difference
Difference in fecal intestinal microbiota composition | day 1-14
Negativization of COVID-PCR at day 14 | day 14
  proportion

CONTACTS AND LOCATIONS:
Overall Officials: Maria M Piskorz, MD, Principal Investigator — Hospital de Clinicas Universidad de Buenos Aires
Locations (1):
- Hospital de Clinicas, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Theisen LL, Erdelmeier CA, Spoden GA, Boukhallouk F, Sausy A, Florin L, Muller CP. Tannins from Hamamelis virginiana bark extract: characterization and improvement of the antiviral efficacy against influenza A virus and human papillomavirus. PLoS One. 2014 Jan 31;9(1):e88062. doi: 10.1371/journal.pone.0088062. eCollection 2014. PMID 24498245
- [Background] Ueda K, Kawabata R, Irie T, Nakai Y, Tohya Y, Sakaguchi T. Inactivation of pathogenic viruses by plant-derived tannins: strong effects of extracts from persimmon (Diospyros kaki) on a broad range of viruses. PLoS One. 2013;8(1):e55343. doi: 10.1371/journal.pone.0055343. Epub 2013 Jan 25. PMID 23372851
- [Background] Zhang L, Cheng YX, Liu AL, Wang HD, Wang YL, Du GH. Antioxidant, anti-inflammatory and anti-influenza properties of components from Chaenomeles speciosa. Molecules. 2010 Nov 22;15(11):8507-17. doi: 10.3390/molecules15118507. PMID 21102377
- [Derived] Molino S, Pisarevsky A, Mingorance FL, Vega P, Stefanolo JP, Repetti J, Luduena G, Pepa P, Olmos JI, Fermepin MR, Uehara T, Villapol S, Savidge T, Treangen T, Viciani E, Castagnetti A, Piskorz MM. Natural tannin extracts supplementation for COVID-19 patients (TanCOVID): a structured summary of a study protocol for a randomized controlled trial. Trials. 2021 Apr 28;22(1):310. doi: 10.1186/s13063-021-05281-x. PMID 33910614